CLINICAL TRIAL: NCT06043856
Title: Translation, Cultural Adaptation and Psychometric Analysis of Urdu Version of Stroke Specific Quality of Life Scale in Stroke Patients
Brief Title: Translation and Psychometric Analysis of the Urdu Version of Stroke Specific Quality of Life Scale
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-UOL-FAHS/1083/2021
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Stroke, Ischemic; Quality of Life
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is a leading cause of adult disability worldwide, ranking as the third major cause of mortality in wealthy nations and the second in developing ones. When adapting a questionnaire for use in a different cultural context, a process called "cross-cultural adaptation" considers linguistic and cultural nuances. Guidelines outline the standard procedure to translate, assess psychometric properties, and culturally adapt questionnaires for new populations.

The Stroke Specific Quality of Life (SS-QOL), designed for self-administration, requires no training. Research indicates its accuracy in assessing stroke victims over the phone, with completion taking 10 to 15 minutes. Scores on the SS-QOL scale correlate with improved functioning. Internal consistency, measured by Cronbach's alpha, ranged from satisfactory to outstanding in stroke patients, indicating good reliability.

This study aims to fill a gap by translating the SS-QOL questionnaire into Urdu, facilitating culturally adapted assessments. Validating scores within the Pakistani population will establish the reliability and effectiveness of the Urdu version, addressing a literature gap in stroke-related quality of life assessments among Urdu speakers in Pakistan. This research aims to provide valuable insights and a comprehensive tool for clinical setups in diverse settings, urban or rural. Introducing a standardized gold standard test will enable healthcare professionals to confidently diagnose and prognose stroke patients. The SS-QOL questionnaire, with its 49 self-report items covering 12 energy-related domains, promises to enhance understanding of stroke's impact on the quality of life among Urdu speakers.

DETAILED DESCRIPTION:
A cross-sectional study was conducted on 147 stroke patients at the Physiotherapy Department of the University of Lahore Teaching Hospital, situated on Defense Road, Lahore. The study spanned nine months following the approval of the research synopsis. Participant selection utilized a non-probability convenient sampling technique. The inclusion criteria comprised stroke-diagnosed patients aged between 35 to 65 years, proficient in verbal Urdu communication. Patients with neurological conditions like Parkinson's disease, Alzheimer's disease, or dementia, as well as unconscious individuals, were excluded. Additionally, patients with musculoskeletal or orthopedic conditions potentially affecting upper and lower extremity functioning were also excluded.

Written informed consent was obtained from all patients, and approval was secured from the Ethics Committee of the University of Lahore. The translated Urdu version of the SS-QOL questionnaire underwent a four-step procedure. Initially, two native Urdu speakers independently translated the SS-QOL into Urdu, with one possessing medical expertise and the other from a non-medical background. Their translations were merged into a single version. This combined version was then translated back into English by two professional translators unfamiliar with the questionnaire and medical terminology to ensure consistent English translation.

A research committee, comprising physiotherapists, an orthopedic surgeon, translators, a language expert, and authors, held a meeting to assess all versions of the SS-QOL for alignment with Urdu cultural nuances and methodological accuracy. After methodological and grammatical analysis, a pre-final SS-QOL version was approved by the committee. Seventy patients confirmed their comprehension of the questions through pilot testing, and their feedback was deliberated upon by the authors. Subsequently, a final Urdu version of the SS-QOL was established.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed stroke patients
* Age between 35 to 65 years 47
* Patients should understand and can verbally communicate in Urdu

Exclusion Criteria:

* Patient with other neurological conditions like parkinson, Alzheimer, Dementia etc
* Unconscious patient
* Patients with musculoskeletal and orthopedic conditions that affect upper and lower extremities function

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosed Stroke Population within range of 35-65 years and possessed the ability to comprehend and communicate verbally in the Urdu language.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Short Form 12 (SF-12) | 1 week
  The SF-12, or Short Form-12, is a widely used self-reported questionnaire used to assess health-related quality of life (HRQOL). It is a shorter version of the SF-36 (Short Form-36), which is a more extensive health survey. The SF-12 is designed to be a concise tool for measuring various aspects of a person's physical and mental health. The SF-12 questionnaire generates two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). These scores provide a way to interpret the overall health-related quality of life of an individual.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Maria Hira, MSPTN, Principal Investigator — University of Lahore; Umair Ahmed, PhD PT, Study Director — University of Lahore; Hafiza Sana Ashraf, MSPT MSK, Study Director — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan